CLINICAL TRIAL: NCT06167616
Title: Infections and Genetic Susceptibility in LADA and Type 2 Diabetes
Brief Title: Infections and Latent Autoimmune Diabetes in Adults
Acronym: LADA
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government); Swedish Council for Working Life and Social Research (Other); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Sofia Carlsson, Associate professor, Karolinska Institutet
Other Study IDs: 2022-00811_1; 2018-03035 (Other Grant/Funding Number: Swedish Research Council); 2018-00337 (Other Grant/Funding Number: FORTE); NNF19OC0057274 (Other Grant/Funding Number: Novo Nordisk Foundation)
Record Dates: First submitted 2023-11-27; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Latent Autoimmune Diabetes in Adults; Type 2 Diabetes
Keywords: Latent Autoimmune Diabetes in Adults; Infections; Diabetes Mellitus; Type 2 diabetes; Case-Control Studies; register study
MeSH Terms: conditions — Latent Autoimmune Diabetes in Adults; Diabetes Mellitus, Type 2; Infections; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- LADA: Classification of LADA based on age ≥35 years at diagnosis, GADA positivity (≥10 U/ml) and C-peptide concentrations of ≥0.2 nmol/L (IMMULITE) or ≥0.3 nmol/L (Cobas).
- Type 2 diabetes: ≥35 years, GADA negative and C-peptide concentrations of >0.60 (IMMULITE)/>0.72 (Cobas) nmol/L.
- Controls: ≥35 years, free of diabetes

SUMMARY:
Infections are proposed risk factors for type 1 diabetes in children. The investigators will examine whether a diagnosis of infectious disease also confers an increased risk of latent autoimmune diabetes in adults.

DETAILED DESCRIPTION:
The investigators will use data from a population-based Swedish case-control study (ESTRID) with incident cases of LADA (n=597) and matched controls (n=2386). History of infectious disease are ascertained through national and regional patient registers. The investigators will estimate adjusted odds ratios (OR) with 95% CI for ≥1 respiratory (any/upper/lower), gastrointestinal, herpetic, other or any infectious disease episode, or separately, for 1 and ≥2 infectious disease episodes, within 0-1, 1-3, 3-5 and 5-10 years before LADA diagnosis/matching. Stratified analyses will be performed based on HLA risk genotypes and GADA levels.

ELIGIBILITY:
Inclusion Criteria:

* 35 years or older, residing in Scania or Uppsala county.

Exclusion Criteria:

* Less than 35 years

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 35 years or older, residing in Scania or Uppsala county.
Sampling Method: Probability Sample
Enrollment: 5048 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
LADA | Up to 10 years
  ≥35 years at diagnosis, GADA positivity (≥10 U/ml) and C-peptide concentrations of ≥0.2 nmol/L (IMMULITE) or ≥0.3 nmol/L (Cobas).

SECONDARY OUTCOMES:
Type 2 diabetes | Up to 10 years
  also ≥35, GADA negative and had C-peptide concentrations of >0.60 (IMMULITE)/>0.72 (Cobas) nmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Carlsson, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institute, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ESTRID website — https://ki.se/en/imm/estrid